CLINICAL TRIAL: NCT00269828
Title: Paclitaxel Poliglumex (CT-2103) vs. Paclitaxel for the Treatment of Women With Chemotherapy-Naïve Advanced Non-Small Cell Lung Cancer (NSCLC) Who Are Performance Status 2.
Brief Title: A Survival Study for Women With Advanced Lung Cancer Who Have Not Previously Received Chemotherapy.
Acronym: PIONEER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGT305; NCT00317824 (obsolete NCT alias)
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: NSCLC
Keywords: Non-small cell lung cancer; NSCLC; PS 2; female; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; paclitaxel poliglumex

INTERVENTIONS:
Drug: paclitaxel
Drug: paclitaxel poliglumex

SUMMARY:
This is a randomized, open-label, multinational, phase III study in women with histologically- or cytologically-confirmed advanced NSCLC who are chemotherapy naïve and have PS 2. Study drug will be administered on day 1 of each 21 day cycle

DETAILED DESCRIPTION:
See Summary

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Histologically- or cytologically-confirmed diagnosis of NSCLC.
3. ECOG performance score of 2.
4. Patients who meet one of the following criteria:

   * Stage IIIB who are not candidates for combined modality therapy (primary radiation therapy or surgery), or
   * Stage IV.
5. Age greater than or equal to 18 years.
6. Adequate bone marrow function
7. Adequate renal function
8. Adequate hepatic function
9. Patients with known brain metastases must have received standard antitumor treatment for their CNS metastases as defined by the site's institutional standards.
10. Patients who have had major surgery must be fully recovered from the surgery.
11. Ability to comply with the visit schedule and assessments required by the protocol.
12. For patients of reproductive potential, commitment to use adequate contraception.
13. Signed approved informed consent, with understanding of study procedures.
14. Agreement to begin study therapy within 8 calendar days after randomization.

Exclusion Criteria:

1. Any intolerance to poly-L-glutamic acid, Poloxamer 188, dibasic sodium phosphate, monobasic sodium phosphate (the excipients of CT-2103).
2. Evidence of small cell carcinoma, carcinoid, or mixed small cell/non-small cell histology.
3. Any prior systemic chemotherapy for the treatment of lung cancer. This includes systemic radiosensitizers used to treat brain metastases and any biologic agent.
4. Concurrent primary malignancies except for carcinoma in situ or non-melanoma skin cancer.
5. Grade 2 or greater neuropathy.
6. Evidence of significant unstable neurological symptoms within the 4 weeks before study randomization. (If unstable neurologic symptoms resulted from brain metastases, patient must meet inclusion criteria number 9).
7. Clinically significant active infection for which active therapy is underway.
8. Investigational therapy within 4 weeks before randomization, unless local requirements are more stringent.
9. Unstable medical conditions including unstable angina or myocardial infarction within the past 6 months before randomization. Patients with evidence of cardiac conduction abnormalities are eligible if their cardiac status is stable.
10. Pregnant women or nursing mothers.
11. Any circumstance at the time of study entry that would preclude completion of the study or the required follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-12; Study Completion 2006-12

PRIMARY OUTCOMES:
The primary objective of this study is to compare the overall survival of female patients randomized to CT-2103 to that of female patients randomized to paclitaxel.

SECONDARY OUTCOMES:
Secondary objectives are to compare the progression-free survival, response rate, disease control, clinical benefit, quality of life, and the safety and tolerability of the treatment arms.

CONTACTS AND LOCATIONS:
Locations (143):
- United States (64):
  - Desert Oasis Cancer Center, Casa Grande, Arizona
  - Arizona Hematology Oncology, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Heritage Physician Group, Oncology, Hot Springs, Arkansas
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Providence St. Joseph Medical Center, Burbank, California
  - Hematology/Oncology Group of Fresno, Inc, Fresno, California
  - Comprehensive Cancer Center-Research Office, Glendale, California
  - Loma Linda University Cancer Institute, Loma Linda, California
  - Pacific Shores Medical Group, Long Beach, California
  - Medical Oncology Care Associates, Orange, California
  - The Cancer Research and Prevention Center, Soquel, California
  - Bethesda Research Center, Boynton Beach, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Florida Wellcare, Inverness, Florida
  - Cancer & Blood Disease Center, Lecanto, Florida
  - Oncology-Hematology Associates of West Broward, Tamarac, Florida
  - Hematology Oncology Speaclist, Tampa, Florida
  - Joliet Oncology Hematology Associates, Ltd., Joliet, Illinois
  - Loyola University Health Systems, Maywood, Illinois
  - Mid-Illinois HEM & ONC Assoc., Normal, Illinois
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Associated Physicians & Surgeons Clinic, Terre Haute, Indiana
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - West Kentucky Hematology & Oncology Group, PSC, Paducah, Kentucky
  - Cabrini Center for Cancer Care, Alexandria, Louisiana
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Troy, Michigan
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - St. Louis Cancer Care Center, Chesterfield, Missouri
  - Columbia Comprehensive Cancer Care Clinics, Columbia, Missouri
  - Bond Clinic, Rolla, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University Siteman Cancer Center Pharmacy, St Louis, Missouri
  - Montana Cancer Specialists, Missoula, Montana
  - Sierra Nevada Oncology Care, Carson City, Nevada
  - Essex Oncology of North Jersey, PA, Belleville, New Jersey
  - Atlanta HEM ONC, Manasquan, New Jersey
  - Oncology and Hematology Specialist, PA, Mountain Lakes, New Jersey
  - San Juan Oncology Association, Farmington, New Mexico
  - Suny Downstate Medical Center, Brooklyn, New York
  - Cancer Treatment Services, Corning, New York
  - Interlakes Foundation, Inc., Rochester, New York
  - Guthrie Clinic, Sayre, New York
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - New York Medical Collegw, Valhalla, New York
  - Alamance Cancer Center, Burlington, North Carolina
  - UNC Chapel Hill Oncology Protocol Office, Chapel Hill, North Carolina
  - Leo Jenkins Cancer Center, Greenville, North Carolina
  - Northwestern Carolina Oncology & Hematology, Hickory, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - University of Cleveland, Cleveland, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Taussig Cancer Center, Cleveland, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Signal Point Hematology/Oncology, Inc., Middletown, Ohio
  - Charleston Hematology Oncology, Charleston, South Carolina
  - The Family Cancer Center, Collierville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
  - JPS Center for Cancer Care, Fort Worth, Texas
  - Columbia Basin HEM/ONC, Kennewick, Washington
- Argentina (8):
  - Sanatorio Parque, Rosario, Santa Fe Province
  - CETEN, Beunos Aires
  - Hospital Privado de Comunidad, Buenos Aires
  - Hospital General de Agudos "Dr Teodoro Alvarez", Buenos Aires
  - Instituto Alexander Fleming, Ciudad de Buenos Aires
  - Instituto Oncologico de Cordoba - IONC, Córdoba
  - LUCEN, Cuidad Autonoma de Buenos Aires
  - ISIS Clinica Especializada, Urquiza
- Bulgaria (8):
  - District Oncology Dispensary, Plovdiv
  - District Oncolodispensary with Impatient sector, Rousse
  - Military Medical Academy, Sofia
  - Regional Oncology Dispensary with Inpatient Secot-Sofia District, Sogia
  - Regional Oncology Dispensary with Inpatient Sector, Varna
  - University Mulitprofile Hospital for Active Treatment "Sveta Marina", Varna
  - University Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
  - Regional Oncology Dispensary with Inpatient sector, Veliko Tarnovo
- Jewish General Hospital, Montreal, Quebec, Canada
- Hungary (10):
  - Erzsebet Juhasz, Budapest
  - University of Debrecen, Pulmonology Clinic, Debreen
  - Hospital for Thoracic Diseases of Csongrad Country, Deszk
  - Pulmonology Institute of Veszprem County, Farkasgyepű
  - Hospital for Pulmonological Diseases of the Bekes County, Gyula
  - Hospital of the Chest Desease of the Hungarian Reformed Church, Mosdós
  - Karolina Hospital, Mosonmagyaróvár
  - Barany County Hospital, Pécs
  - Erzsebet Hospital, Sopron
  - Sanatorium for Pulmonological Diseases, Törökbálint
- Mexico (12):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes, Aguascalientes
  - CIMA Chihuahua, Chihuahua City, Chih
  - Hospital General, Durango, Durango
  - Instituto Estatal de Cancerologia "Dr. Arturo Beltran Ortega", Acapulco de Juárez, Guerrero
  - Hospital Dr. Angel Leano, Zapopan, Jalisco
  - Hospital Star Medica Morelina, Morelia, Michoacán
  - Monterrey International Research Center, Monterrey, N.L.
  - Centro Estatal de Canceologia, Jalapa, Veracruz
  - Centro Anticanceroso de la Cruz Roja Mexicana de Merida, Mérida, Yucatán
  - Centro Estatal de Cancerologia, Chihuahua City
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
  - Hospital General Regional, Veracruz
- Poland (9):
  - Kujawsko-Pomorskie Centrum Pulmunologii, Bydgoszcz
  - Krakowski Szpital Specjelistyczny, Kawkow
  - Centrum Onkologii Ziemii Lubelskiej, Lublin
  - Zaklad Opieki Zdrowotnej Ministerstaw Spraw Wewnetrznych i Administraeji, Olsztyn
  - Mazowleckie Centrum leczenia Chorob Pluc i Gruzlicy, Otwock
  - Wielkopolskie Centrum Chorob Pluc i Gruzlicy, Samodzielmy Publiczny ZOZ, Poznan
  - SPSK nr l im. Przemienienia AM w Poznaniu, Poznan
  - MSc Grezegorz Jedrejezak, Wroclaw
  - Dolnoslaskie Centrum Chorob Pluc ul. Grabiszynska 105, Wroclaw
- Romania (7):
  - Institutul Oncologie - Clinic de Oncologie Medicala, Bucharest
  - Prof. Dr. Al. Trestioreanu Institute of Oncology, Bucharest
  - "Prof. Dr. I. Chiricuta" Institute of Oncology, Cluj-Napoca
  - Emergency Clinical County Hospital, Craiova
  - Oradea Clinical County Hospital, Oradea
  - Clinical County Hospital, Sibiu
  - Timisoara Emergency Clinical Municipal Hospital, Timișoara
- Russia (13):
  - Chelyabinsk Regional Oncology Center, Chelyabinsk
  - Krasnodar City Oncology Center, Krasnodar
  - Moscow Oncology Clinical Dispensary #1, Moscow
  - SI Russian Oncological Scientific Center after N.N. Blokhim RAMS, Moscow
  - SI Russian Oncological Scientific Center after N.N. Blokhin RAMS, Moscow
  - Centeral ClinicalHospital of the President o the Russian Federation, Moscow
  - Moscow Municpal Oncology Hospital #62, Moscow Region
  - Omsk Regional Oncology Center, Omsk
  - Orenburg Regional Oncology Clinical Center, Orenburg
  - Lenigrad Regional Oncology Center, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - St. Petersbrug State Medical Pavlov University, Saint Petersburg
  - St. Petersburg City Clinical Oncology Center, Saint Petersburg
- Ukraine (7):
  - Donetsk Regional Antineoplastic Center, Donetsk
  - Ivano-Frankovsk Regional Oncology Center, Ivano-Frankovsk Medical University, Ivano-Frankivsk
  - Instiute of Oncology under AMS of Ukraine, Kiev
  - Volyn Regional Oncology Dispensary, Lutsk
  - Uzhgorod National University, Regional Clinical Oncology Dispensary, Uzhhorod
  - Vinnitsa State Medical University, Vynnytsya
  - Zaporizhzhya Regional Oncology Dispensary, Zaprizhzhya
- United Kingdom (4):
  - The Royal Bournemouth Hospital, Bournemouth
  - Oncology Pharmacy, London
  - Wythenshaw Hospital, Pharmacy Department, Manchester
  - Southhampton General Hospital, Southhampton